CLINICAL TRIAL: NCT03091595
Title: A Single-center, Randomized, Open-label, Two-arm Study to Evaluate the Ovarian Function Inhibition of a Monophasic Combined Oral Contraceptive (COC) Containing 15 mg Estetrol (E4) and 3 mg Drospirenone (DRSP) and a Monophasic COC Containing 20mcg Ethinylestradiol (EE)/3 mg DRSP (YAZ®), Administered Orally Once Daily in a 24/4 Day Regimen for Three Consecutive Cycles
Brief Title: E4/DRSP Ovarian Function Inhibition Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Estetra (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MIT-Es0001-C202; 2016-004267-40 (EudraCT Number)
Record Dates: First submitted 2017-03-21; First posted 2017-03-27 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-04

CONDITIONS: Prevention of Pregnancy
MeSH Terms: interventions — drospirenone; drospirenone and ethinyl estradiol combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 15 mg E4/3 mg DRSP (Experimental): 15 mg E4 combined with 3 mg DRSP administered in a 24/4-day regimen. One tablet per day orally for 3 treatment cycles.
  Interventions: Drug: 15 mg E4/3 mg DRSP
- 20 mcg EE/3 mg DRSP (Active Comparator): 20 mcg EE combined with 3 mg DRSP administered in a 24/4-day regimen. One tablet per day orally for 3 treatment cycles.
  Interventions: Drug: 20 mcg EE/3 mg DRSP

INTERVENTIONS:
Drug: 15 mg E4/3 mg DRSP — 15 mg E4/3 mg DRSP combined tablets will be administered orally once daily in a 24/4 day regimen for three consecutive cycles
  Other Names: 15 mg estetrol combined with 3 mg drospirenone
  Arms: 15 mg E4/3 mg DRSP
Drug: 20 mcg EE/3 mg DRSP — 20 mcg EE/3 mg DRSP combined tablets will be administered orally once daily in a 24/4 day regimen for three consecutive cycles
  Other Names: 20 mcg ethinylestradiol combined with 3 mg drospirenone (Yaz)
  Arms: 20 mcg EE/3 mg DRSP

SUMMARY:
A combined oral contraceptive (COC) containing 15 mg E4 and 3 mg DRSP administered for 24 days followed by 4 placebo tablets, is being evaluated for further development. This study will investigate the effect of this COC on ovarian function inhibition, levels of serum luteinizing hormone (LH), follicle-stimulating hormone (FSH), estradiol (E2) and progesterone during 3 treatment cycles in comparison with the reference COC 20 mcg EE/3 mg DRSP.

ELIGIBILITY:
Inclusion Criteria:

* Overtly healthy female subjects, as determined by medical history, physical examination including breast examination, gynecological examination (including cervical smear [Pap smear]), vital signs, ECG, echocardiogram, and laboratory tests.
* Negative pregnancy test at subject screening.
* Women who ovulate in the Pre-Treatment Cycle.
* Willing to use a non-hormonal method of contraception (e.g. condom) during the wash-out period, Pre-Treatment Cycle and Post-Treatment Cycle.
* BMI between 18.0 and 35.0 kg/m², inclusive, at time of Screening.
* Able to fulfill the requirements of the protocol and have indicated a willingness to participate in the study by providing written informed consent form (ICF).

Exclusion Criteria:

* Irregular menstrual cycle.
* Amenorrhea or abnormal uterine bleeding.
* Clinically relevant abnormal laboratory result at Screening.
* Clinically significant abnormalities of the uterus and/or ovaries detected by examination and/or ultrasound.
* Known hypersensitivity to any of the investigational or reference product ingredients.
* Intention to become pregnant during the course of the study.
* Pregnancy during accurate hormonal contraceptive use in the past.
* Dyslipoproteinemia requiring active treatment with antilipidemic agent.
* Diabetes mellitus with vascular involvement (nephropathy, retinopathy, neuropathy, other) or diabetes mellitus of more than 20-year duration.
* Any arterial hypertension.
* Any condition associated with an increased risk of venous thromboembolism and/or arterial thromboembolism.
* Complicated valvular heart disease.
* History of pregnancy-related cardiomyopathy or moderately or severely impaired cardiac function.
* Systemic lupus erythematosus.
* Presence or history of migraine with aura.
* Abnormal Papanicolaou (PAP) smear result.
* Presence of an undiagnosed breast mass.
* Current symptomatic gallbladder disease.
* History of COC-related cholestasis.
* Presence or history of severe hepatic disease.
* Presence or history of pancreatitis if associated with hypertriglyceridemia.
* Porphyria.
* Presence or history of hepatocellular adenoma or malignant liver tumors.
* Renal impairment.
* Hyperkaliemia or presence of conditions that predispose to hyperkaliemia.
* Presence or history of hormone-related malignancy.
* History of non-hormone-related malignancy within 5 years before Screening. Subjects with a non-melanoma skin cancer are allowed in the study.
* Use of drugs potentially triggering interactions with COCs.
* History of alcohol or drug abuse.
* Any prior procedure, disease or condition that could result in altered absorption, excessive accumulation, impaired metabolism, or altered excretion of the investigational product.
* Uncontrolled thyroid disorders.
* Have received an investigational drug within the last 2 cycles prior to start of Pre-Treatment Cycle. Subjects who participated in an oral contraceptive clinical study, using Food and Drug Administration (FDA)/European Union (EU) approved active ingredients, may start the Pre-Treatment Cycle one cycle after last medication intake of the preceding study.
* Sponsor, contract research organization (CRO) or PI's site personnel directly affiliated with this study.
* Is judged by the PI to be unsuitable for any reason.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 82 (Actual)
Dates: Start 2017-02-07 (Actual); Primary Completion 2018-06-08 (Actual); Study Completion 2018-06-08 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects with ovarian inhibition at treatment Cycle 1 | All assessments will be performed once every 3 days starting treatment Cycle 1 Day 3 (± 1 day) until Day 27 (± 1 day) (one treatment cycle = 28 days).
  Ovarian inhibition will be assessed by rating the suppression of ovaries using the Hoogland score. This score is based on:
  * the follicular size assessed by transvaginal ultrasound (TVUS)
  * endogenous hormone levels: serum E2, and serum progesterone.
Proportion of subjects with ovarian inhibition at treatment Cycle 3 | All assessments will be performed once every 3 days starting treatment Cycle 3 Day 3 (± 1 day) until Day 27 (± 1 day) (one treatment cycle = 28 days).
  Ovarian inhibition will be assessed by rating the suppression of ovaries using the Hoogland score. This score is based on:
  * the follicular size assessed by TVUS
  * endogenous hormone levels: serum E2, and serum progesterone.

SECONDARY OUTCOMES:
Serum level of luteinizing hormone (LH) | On cycle Day 3, 6, 9, 12, 15, 18, 21, 24, 27 at treatment Cycle 1 and treatment Cycle 3 and on cycle Day 3 of the Treatment Cycle 2 (each treatment cycle = 28 days)
  Blood samples will be taken at regular time points defined in the time frame.
Serum level of follicle stimulating hormone (FSH) | On cycle Day 3, 6, 9, 12, 15, 18, 21, 24, 27 at treatment Cycle 1 and treatment Cycle 3 and on cycle Day 3 of the Treatment Cycle 2 (each treatment cycle = 28 days)
  Blood samples will be taken at regular time points defined in the time frame.
Serum level of estradiol (E2) | On cycle Day 3, 6, 9, 12, 15, 18, 21, 24, 27 at treatment Cycle 1 and treatment Cycle 3 and on cycle Day 3 of the Treatment Cycle 2 (each treatment cycle = 28 days)
  Blood samples will be taken at regular time points defined in the time frame.
Serum level of progesterone (P) | On cycle Day 3, 6, 9, 12, 15, 18, 21, 24, 27 at treatment Cycle 1 and treatment Cycle 3 and on cycle Day 3 of the Treatment Cycle 2 (each treatment cycle = 28 days)
  Blood samples will be taken at regular time points defined in the time frame.
Maximum endometrial thickness | From Baseline (study day 1), through 3 treatment cycles and up to Cycle Day 36 (±1) of the Post-Treatment Cycle (study day 120 (±1)) (each treatment cycle = 28 days)
  Endometrial thickness will be measured using transvaginal ultrasound (TVUS). Maximum endometrial thickness was defined as the largest endometrial thickness during a cycle.
Mean diameter of the largest follicle | Day 3 to Day 24 of Post-Treatment Cycle
  Follicular size will be measured using TVUS.
Number of participants who experience at least one Treatment-Emergent Adverse Event (TEAE) | Day 1 to Follow-Up Visit (+ 30 days)
Number of participants who experience pregnancy during treatment | Cycle 1 Day 1 to Follow-Up Visit (+ 30 days) (each treatment cycle = 28 days)
Number of participants who experience a clinically significant change in physical examination results | Day 1 to End of Follow-Up Visit (+ 30 Days)
Number of participants who experience a clinically significant change in gynecological examination results | Day 1 to End of Follow-Up Visit (+ 30 Days)
Number of participants who experience a clinically significant change in clinical laboratory results | Day 1 to End of Follow-Up Visit (+ 30 Days)
Number of participants who experience a clinically significant change in electrocardiogram (ECG) results | Day 1 to End of Cycle 3 (Day 28) (each treatment cycle = 28 days)
Number of participants who experience a clinically significant change in echocardiogram results | Day 1 to End of Cycle 3 (Day 28) (each treatment cycle = 28 days)
Change from Baseline in diastolic blood pressure | From Baseline (study day 1), through 3 treatment cycles and up to Cycle Day 36 (±1) of the Post-Treatment Cycle (study day 120 (±1)) (each treatment cycle = 28 days)
Change from Baseline in systolic blood pressure | From Baseline (study day 1), through 3 treatment cycles and up to Cycle Day 36 (±1) of the Post-Treatment Cycle (study day 120 (±1)) (each treatment cycle = 28 days)
Change from Baseline in pulse rate | From Baseline (study day 1), through 3 treatment cycles and up to Cycle Day 36 (±1) of the Post-Treatment Cycle (study day 120 (±1)) (each treatment cycle = 28 days)

CONTACTS AND LOCATIONS:
Overall Officials: Christine Klipping, Principal Investigator — Dinox BV
Locations (1):
- Dinox BV, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Trial results were released to public view on the EudraCT (EudraCT Number: 2016-004267-40). — https://www.clinicaltrialsregister.eu/ctr-search/trial/2016-004267-40/results